CLINICAL TRIAL: NCT04026841
Title: The Efficacy of PD-1 Antibody Sintilimab on Early-stage Multiple Primary Lung Cancer With Ground Glass Density: A Prospective Interventional Two-stage Simon Design Phase II Study.
Brief Title: The Efficacy of PD-1 Antibody Sintilimab on Early-stage Multiple Primary Lung Cancer With Ground Glass Density.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCTC1901
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Multiple Primary Lung Cancers
Keywords: ground-glass nodule; ground-glass density

STUDY DESIGN:
Intervention Model Description: Clinical trials with a single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 Antibody Sintilimab (Experimental): Patients receive the treatment of PD-1 antibody Sintilimab
  Interventions: Drug: PD-1 antibody Sintilimab

INTERVENTIONS:
Drug: PD-1 antibody Sintilimab — Patients in experimental group receive the treatment of PD-1 antibody Sintilimab

SUMMARY:
A single-center,prospective interventional study to explore the efficacy of PD-1 antibody Sintilimab on early-stage multiple primary lung cancer patients with ground-glass nodules in CT scan.

DETAILED DESCRIPTION:
This study is a single-center,prospective interventional clinical study, all subjects enrolled are multiple primary lung cancer patients with ground-glass density in CT scan.The samples plan for the study was 36 cases.The enrolled patients will receive intravenous infusion of Sintilimab 200mg every 3 weeks up to 4 cycles, and the efficacy will be evaluated after cycle 2 and 4 using RECIST criteria (version 1.1 ).

ELIGIBILITY:
Inclusion Criteria:

* Two or more ground-glass lesions (pure ground glass or partially solid) presented in the CT scan of lung that cannot be operated simultaneously
* There was at least one lung cancer lesion with a diameter of 1-3cm confirmed pathologically or by multidisciplinary team.
* Excluding lymph nodes and distant metastasis through imaging
* ECOG PS 0-1
* Vital organ functions meet the following requirements: 1)The absolute count of neutrophils ≥1.5×109/L 2)Platelet ≥90×109/L 3)Hemoglobin ≥9g/dL 4)Serum albumin ≥3g/dL 5)Thyroid stimulating hormone (TSH) ≤ULN (if abnormal, T3 and T4 levels should be examined at the same time; if T3 and T4 levels are normal, they can be included in the group) 6)Bilirubin ≤ULN 7)ALT and AST≤1.5 ULN 8)AKP≤ 2.5ULN or less 9)Serum creatinine ≤1.5 ULN or creatinine clearance ≥60mL/min
* Subjects volunteered to participate in this study and signed informed consent, with good compliance.

Exclusion Criteria:

* Non-calcified lesions with diameter more than 3mm are presented
* The presence of any active autoimmune diseases or a history of autoimmune diseases
* Those who have used other drugs in clinical study within 4 weeks before the first time of drug use
* Severe allergic reaction to monoclonal antibody
* Heart clinical symptoms or diseases are not well controlled
* Subjects with congenital or acquired immune deficiency (such as HIV infection) or active hepatitis
* According to the researcher's judgment, the subjects have other factors that may lead to the forced termination of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
ORR of target lesions. | 3 months
  The objective response rate will be evaluated after 4 courses of treatment

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 months
  The safty of PD-1 Antibody Sintilimab

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Department of Thoracic Surgery and Oncology, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China